CLINICAL TRIAL: NCT02823158
Title: A Prospective Randomized Controlled Trial of Bilateral Pallidal Stimulation in Patients With Advanced Parkinson's Disease With Motor Complications and Relative or Absolute Contraindications for Subthalamic Stimulation
Brief Title: Bilateral Pallidal Stimulation in Patients With Advanced Parkinson's Disease-LATESTIM
Acronym: LATESTIM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-000334
Record Dates: First submitted 2016-04-18; First posted 2016-07-06 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Central Nervous System Disease; Basal Ganglia Disease; Movement Disorders; Neurodegenerative Disorders; Parkinson Disease
Keywords: Parkinson Disease; Morbus Parkinson; Basal Ganglia; Pallidal Stimulation
MeSH Terms: conditions — Central Nervous System Diseases; Basal Ganglia Diseases; Movement Disorders; Neurodegenerative Diseases; Parkinson Disease | interventions — Deep Brain Stimulation

ARMS (2):
- GPi DBS and best medical treatment (Experimental)
  Interventions: Procedure: Deep brain stimulation (DBS) of Globus Pallidus internus (GPi) and Best medical treatment (BMT); Procedure: Best medical treatment
- Best medical treatment (Active Comparator)
  Interventions: Procedure: Best medical treatment

INTERVENTIONS:
Procedure: Deep brain stimulation (DBS) of Globus Pallidus internus (GPi) and Best medical treatment (BMT) — Patients in the GPi group will be implanted with DBS-electrodes within 6 weeks after randomisation. The stimulation parameters and the medical treatment are adjusted for optimal control of motor and non-motor signs and symptoms according to published guidelines using a specified algorithm. The stimulation parameters are recorded at the beginning and at the end of each post-surgical assessment.
  Best medical treatment is applied in combination with GPi-DBS.
  Other Names: Bilateral pallidal stimulation; Deep brain stimulation
  Arms: GPi DBS and best medical treatment
Procedure: Best medical treatment — Patients will receive optimized medical treatment according to published evidence based guidelines.

SUMMARY:
Deep brain stimulation (DBS) is an established treatment for advanced complicated Parkinson's disease (PD). Several controlled randomized studies have given proof of an advantage for operated patients as compared to medically treated patients in terms of motor outcome, activities of daily living and health status. However these studies have addressed mostly stimulation of the subthalamic nucleus (STN). GPi stimulation has not been compared to best medical treatment (BMT) in a prospective randomized controlled trial in patients with complicated PD who are not good candidates for STN stimulation. The investigators aim assessing GPi-DBS in patients with PD who have contraindications for STN-DBS.

DETAILED DESCRIPTION:
The indication and excellent therapeutic effects of STN stimulation have been sufficiently proven in advanced PD, and the contraindications for this treatment are rather well established. Also, the observation that patients fulfilling the "STN-profile" but who had been operated for pallidal DBS and lost part of the treatment's benefit over time, improved when stimulated later in the STN (instead of the GPi) shows that patients qualifying for STN-DBS do not have as good a result with GPi-DBS.

GPi stimulation may be used in patients who do not qualify for STN stimulation. Especially postural instability, age over 70 years, and mild to moderate cognitive deficits are commonly considered to be exclusion criteria for STN stimulation but not for GPi stimulation. Therefore, the investigators propose a prospective randomized controlled trial of GPi stimulation in patients with PD and motor complications who have relative or absolute contraindications for STN stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease according to the UKBB criteria, with the exception that familial forms of otherwise typical parkinsonian syndromes may also be included
* motor complications of dopaminergic medication (dyskinesia or motor fluctuations or both) that are at least moderately bothersome to the patient [on a scale of 5 possible levels: not at all / mildly / moderately / severely / extremely bothersome]
* Presence of at least one of the following absolute exclusion criteria for STN stimulation:

  * Mattis dementia rating scale <130 points
  * postural instability of >1 in the item of MDS-UPDRS III [item #12] "on" medication
  * less than 30% improvement of axial score in the acute levodopa challenge test [axial score =sum of items 3.1, 3.9, 3.10, 3.12, 3.13 of the MDS UPDRS III]
* or presence of at least two of the following relative exclusion criteria for STN stimulation:

  * age > 70 years
  * Mattis dementia rating scale <134 points
  * gait freezing "on" medication
  * dysarthria of > 2 in the item of the MDS-UPDRS III [item #3.1]
  * less than 50% improvement of axial score in the acute levodopa challenge test [axial score = sum of items 3.1, 3.9, 3.10, 3.12, 3.13 of the MDS UPDRS III]
  * Starkstein apathy score of ≥14
* Complete baseline PDQ-39-SI and patient diary available
* written informed consent

Exclusion Criteria:

* Age > 85 years
* surgical or medical contraindications
* abnormalities on brain MRI that preclude the implantation of electrodes into the GPi
* contraindication for 3T MRI (baseline imaging)
* severe medical illness that is likely to hamper the benefit of DBS
* severe personality disorder that may interfere with optimization of DBS
* dementia according to DSM-V and MMSE < 20
* ongoing psychosis (except pseudohallucinations)
* ongoing major depression (BDI-II > 23) or depression of any severity with suicidal ideation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Difference of change of the score of the Parkinson's disease questionnaire 39 (PDQ-39-SI) from baseline to follow-up between the two treatment groups. | Baseline and 5 months +/- 1 month
Difference of change in number of hours per day spent in motor "on" without troublesome dyskinesia from baseline to follow-up between the two treatment groups. | Baseline and 5 months +/- 1 month

SECONDARY OUTCOMES:
Difference of change of the score of the MDS-UPDRS part III (Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale, part III) from baseline to follow up between the two trial groups. | Baseline and 5 months +/- 1 month
Difference of change of the score of the MDS-UPDRS part IV (Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale, part IV) (MDS-UPDRS) from baseline to follow up between the two trial groups. | Baseline and 5 months +/- 1 month
Difference of change in number of hours per day spent in motor "on" with troublesome dyskinesia from baseline to follow-up between the two treatment groups. | 5 months +/- 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schüpbach, PD Dr. med, Principal Investigator — Inselspital University Hospital Bern; Ines Debove, Dr. med, Principal Investigator — Inselspital University Hospital Bern
Locations (1):
- Inselspital University Hospital Bern, Bern, Switzerland